CLINICAL TRIAL: NCT06069765
Title: Trunk and Upper Extremities Program Effect in Decreasing Compensation Patterns in Unilateral Cerebral Palsy Children: Randomized Control Trial
Brief Title: Trunk and Upper Extremities Program Effect in Decreasing Compensation Patterns in Unilateral Cerebral Palsy Children
Acronym: TUPEX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio Aspace Catalunya (Other)
Collaborators: Universitat Internacional de Catalunya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TrunkUpperExtremityPrograma
Record Dates: First submitted 2023-09-19; First posted 2023-10-06 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy Infantile; Chronic Pain; Upper Extremity Dysfunction
Keywords: compensation patterns; unilateral cerebral palsy
MeSH Terms: conditions — Cerebral Palsy; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: One member of the research team responsible for carrying out the evaluations of the dependent variables and the collection of data carried out by the participant himself and/or his families, will remain blinded to the assignment of the participants to the study groups.
  In this sense, it is worth saying that the person responsible for carrying out the evaluations will do so only for the main variable, that is to say, he will be the one who will carry out the registration of the compensatory movements of the proximal part of the upper limb and trunk through the DLC . The secondary response variables are evaluated through self-administered scales and this same evaluator will be in charge of collecting the data provided by the families.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard group (No Intervention): Children in this group will continue with their daily activities such as conventional physiotherapy and occupational therapy, even psychology, and their physical activities such as swimming or playing football.
- TUPEX group (Experimental): Children in this group will continue with their daily activities and will add the TUPEX program during 8 weeks.
  Interventions: Other: TUPEX

INTERVENTIONS:
Other: TUPEX — This program contains exercises with their own body weight or with Thera-bands for gaining strength in their shoulder and trunk muscles. It contains some progression exercise if needed.
  Each session can last between 20 and 30 minutes. Children have to do each session three times a week during 8 weeks.
  Arms: TUPEX group

SUMMARY:
The goal of this clinical trial is to test the effectiveness of a trunk and upper extremities exercise program. The main questions it aims to answer are:

Whether the program decreases compensation patterns in unilateral cerebral palsy children Whether the program decreases pain in unilateral cerebral palsy children Whether the program improves bimanual ability in unilateral cerebral palsy children Participants will undertake and 8-week program exercise at home If there is a comparison group: Researchers will compare with the control group to see if this program decreases compensation patterns.

DETAILED DESCRIPTION:
Children in control group will continue with their daily activities. Children in experimental group, apart from their daily activities, will undertake an 8-week program exercise at home for strengthening the trunk and the proximal part of both upper extremities. It contains 3 progressions that can be applied if needed.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral cerebral palsy diagnostic
* Level I or II of the Manual Ability Scale Classification

Exclusion Criteria:

* Have received any intervention with botulinum toxin or shock waves in the previous six months or have them scheduled during the intervention
* Are undergoing treatment with intensive therapies.
* To have known alteration in the hips
* Have very serious attention or comprehension difficulties that prevent them from following instructions.
* Suffer uncontrolled epilepsies
* Suffer from severe visual problems.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Rate of variance of the Compensation patterns | 8 weeks
  DeepLabCut (DLC) (Artificial Intelligence). Calculate the kinematic difference of the body marks during the activities

SECONDARY OUTCOMES:
Intensity of pain | 8 weeks
  Face Pain Scale - Revised (FPS-R). The face marked is compared before and after the treatment. 0 is the minimum scores, meaning no pain, and 10 is the maximum score, meaning really severe pain.
Location of pain | 8 weeks
  In the Body Diagram. The location of the pain is compared before and after the treatment
Bimanual ability | 8 weeks
  Children Hand-Use Experience Questionaire 2.0 (CHEQ 2.0). Whether they are more capable of doing more bimanual activities or not. The maximum score in each question is 100 and the minimum is 0. 100 means children use their hands like the neurotypical children, and 0 means they can't use the affected hand at all.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Biedermann, Study Chair — Aspace Catalunya

IPD SHARING:
Plan to Share IPD: Yes
The results could be submitted for publication in Clinical Rehabilitation, Therapeutic Advances in Chronic Disease, Acta Pediatrics or in Developmental Medicine & Child Neurology (DMCN).
  It is also planned to disseminate the knowledge obtained to different associations in the field of physiotherapy in pediatrics such as the Spanish Association of Intervention in the Early Childhood (AEIPI) and the Spanish Pediatric Association (AEP) or Association of Infantile Hemiparesis.
  Regarding the presentation at congresses, it is planned to present the results of this study at the annual congress of the European Academy of Childhood Disability, that of the Spanish Society of Child Rehabilitation or the National Congress of Rehabilitation.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The research group expects to start sharing results at the end of 2024
Access Criteria: Open

REFERENCES:
- [Result] Abd-Elfattah HM, Aly SM. Effect of Core Stability Exercises on Hand Functions in Children With Hemiplegic Cerebral Palsy. Ann Rehabil Med. 2021 Feb;45(1):71-78. doi: 10.5535/arm.20124. Epub 2021 Feb 9. PMID 33557483
- [Result] Mckinnon CT, Meehan EM, Harvey AR, Antolovich GC, Morgan PE. Prevalence and characteristics of pain in children and young adults with cerebral palsy: a systematic review. Dev Med Child Neurol. 2019 Mar;61(3):305-314. doi: 10.1111/dmcn.14111. Epub 2018 Dec 3. PMID 30508221
- [Result] Brochard S, Lempereur M, Mao L, Remy-Neris O. The role of the scapulo-thoracic and gleno-humeral joints in upper-limb motion in children with hemiplegic cerebral palsy. Clin Biomech (Bristol). 2012 Aug;27(7):652-60. doi: 10.1016/j.clinbiomech.2012.04.001. Epub 2012 May 2. PMID 22560625
- [Result] Francisco-Martinez C, Prado-Olivarez J, Padilla-Medina JA, Diaz-Carmona J, Perez-Pinal FJ, Barranco-Gutierrez AI, Martinez-Nolasco JJ. Upper Limb Movement Measurement Systems for Cerebral Palsy: A Systematic Literature Review. Sensors (Basel). 2021 Nov 26;21(23):7884. doi: 10.3390/s21237884. PMID 34883885
- [Result] Jackman M, Sakzewski L, Morgan C, Boyd RN, Brennan SE, Langdon K, Toovey RAM, Greaves S, Thorley M, Novak I. Interventions to improve physical function for children and young people with cerebral palsy: international clinical practice guideline. Dev Med Child Neurol. 2022 May;64(5):536-549. doi: 10.1111/dmcn.15055. Epub 2021 Sep 21. PMID 34549424
- [Result] Novak I. Evidence-based diagnosis, health care, and rehabilitation for children with cerebral palsy. J Child Neurol. 2014 Aug;29(8):1141-56. doi: 10.1177/0883073814535503. Epub 2014 Jun 22. PMID 24958005